CLINICAL TRIAL: NCT02798289
Title: A Single Arm, Multicenter, Open-Label Study Designed to Evaluate Acute Tear Production Following Single Use of the Oculeve Intranasal Neurostimulator
Brief Title: Acute Tear Production Following Single Use of the Oculeve Intranasal Neurostimulator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oculeve, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OCUN-014
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Results first posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-09

CONDITIONS: Dry Eye Syndrome; Keratoconjunctivitis Sicca
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active - Device (Experimental): The Oculeve Intranasal Neurostimulator will be administered once to induce aqueous tear production once following study enrollment.
  Interventions: Device: Oculeve Intranasal Neurostimulator

INTERVENTIONS:
Device: Oculeve Intranasal Neurostimulator — Neurostimulation device

SUMMARY:
The primary objective of this study is to evaluate acute tear production as measured by tear meniscus height (TMH) captured by optical coherence tomography (OCT) after single use of the Oculeve Intranasal Neurostimulator (OIN) in participants with dry eye.

DETAILED DESCRIPTION:
This is a prospective, single-arm, multicenter, open-label clinical trial in which participants will use the OIN once following study enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with dry eye disease
* Literate, able to speak English or Spanish, and able to complete questionnaires independently
* Willing to sign the informed consent and deemed capable of complying with the requirements of the study protocol

Exclusion Criteria:

* Chronic or recurrent epistaxis, coagulation disorders or other conditions that, in the opinion of the investigator, may lead to clinically significant increased bleeding
* Nasal or sinus surgery (including history of application of nasal cautery) or significant trauma
* Cardiac demand pacemaker, implanted defibrillator or other implanted electronic device
* Corneal transplant in either or both eyes
* Participation in any clinical trial with a new active substance or a new device within 30 days of the Screening Visit
* Women who are pregnant, planning a pregnancy, or nursing at the Screening Visit

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Friedman, MD, Study Director — Mid-Peninsula Ophthalmology Medical Group
Locations (2):
- United States (2):
  - Sall Research Medical Center, Artesia, California
  - Aesthetic Eyecare Institute, Newport Beach, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Active - Device: The Oculeve Intranasal Neurostimulator will be administered once to induce aqueous tear production following study enrollment. Oculeve Intranasal Neurostimulator: Neurostimulation device
Period: Overall Study
Arm/Group | Active - Device
Started | 55
Completed | 55
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Active - Device
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 37
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Tear Meniscus Height Captured by Optical Coherence Tomography
Description: Tear meniscus Height was measured before and after stimulation with Oculeve Intranasal Neurostimulator using Optical Coherence Tomography.
Time Frame: Day 1
Population: Safety population included all subjects who received device intervention.
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Active - Device
Number analyzed (Participants) | 55
µm
  Pre-stimulation TMH | 238.4 (16.7)
  Post-stimulation TMH | 634.9 (60.8)

ADVERSE EVENTS:
Time Frame: Day 0 to Day 22
Groups:
- Active - Device: The Oculeve Intranasal Neurostimulator will be administered once to induce aqueous tear production once following study enrollment. Oculeve Intranasal Neurostimulator: Neurostimulation device
Arm/Group | Active - Device
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The data provided by this clinical trial, and all related information and any materials containing such data and information, are the exclusive property of Oculeve and are confidential to Oculeve. The investigator or other study-related personnel may not disclose to anyone or use any data, information, or materials related to this clinical trial without the express written consent of Oculeve.